CLINICAL TRIAL: NCT06150664
Title: A Phase 1, Open-Label, Multiple-Ascending Dose Study of the Safety and Tolerability of CTX-8371 in Patients With Advanced Malignancies
Brief Title: A Phase 1 of CTX-8371 in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Compass Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTX-8371-001
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Triple Negative Breast Cancer; Hodgkin Lymphoma; Head and Neck Squamous Cell Carcinoma; Malignant Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Hodgkin Disease; Squamous Cell Carcinoma of Head and Neck; Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort 1 (Experimental): Escalating doses of CTX-8371
  Interventions: Drug: CTX-8371
- Dose Expansion Cohort 2 (Experimental): Two CTX-8371 dose groups (3.0 mg/kg and 10.0 mg/kg) in two tumor type subgroups (NSCLC and TNBC)
  Interventions: Drug: CTX-8371

INTERVENTIONS:
Drug: CTX-8371 — Intravenous (IV) infusion every two weeks.

SUMMARY:
This is a Phase 1, open-label, first-in-human study of CTX-8371 administered as a monotherapy in patients with metastatic or locally advanced malignancies. The study will be conducted in 2 cohorts: Dose Escalation and Dose Expansion.

DETAILED DESCRIPTION:
This Phase 1, open-label, first-in-human study will evaluate the safety, tolerability, immunogenicity, and pharmacokinetic profile of CTX-8371 monotherapy. Preliminary anti-tumor activity of CTX-8371 will also be assessed. The study will be conducted in 2 cohorts: Dose escalation and Dose expansion. The Dose Escalation Cohort will utilize a 3+3 design to evaluate five dose levels (0.1-10.0 mg/kg) of CTX-8371 given as an IV infusion once every 2 weeks. Patients in the Dose Expansion Cohort will receive CTX-8371 as an IV infusion at 3.0 mg/kg or 10.0 mg/kg at a 1:1 allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patients must have a histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic disease that is relapsed/refractory to standard therapy or for which no effective standard therapy is available, including

   1. Malignant Melanoma (MM)

      * Patients who have progressed after a minimum of 2 doses of a PD-1/PD-L1 treatment. Study enrollment (C1D1) must be within 12 weeks of the last dose of the anti-PD-1/PD-L1 blocking antibody
      * Patients must have had prior testing for BRAF V600 mutations. Patients with BRAF V600 activating mutation must have received prior therapy with a BRAF/MEK inhibitor
      * Uveal and mucosal melanoma are excluded
   2. Head and Neck squamous cell carcinoma (HNSCC)

      * HNSCC of oral cavity, oropharynx, hypopharynx, or larynx
      * Patients who have progressed after a minimum of 2 doses of a PD-1/PD-L1 treatment. Study enrollment (C1D1) must be within 12 weeks of the last dose of the anti-PD-1/PD-L1 blocking antibody
      * Patients must have received prior treatment with platinum-based chemotherapy
   3. Non-Small Cell Lung Cancer (NSCLC)

      * Patients who have progressed after a minimum of 2 doses of a PD-1/PD-L1 treatment. Study enrollment (C1D1) must be within 12 weeks of the last dose of the anti-PD-1/PD-L1 blocking antibody
      * Patients must have received prior treatment with platinum-based chemotherapy
   4. Triple Negative Breast Cancer (TNBC)

      * ER/PR and HER2 status should be defined by ASCO/CAP guidelines (JCO Allison et al 2020)
      * Patients with HER2-low cancers (HER2 IHC 1+ or 2+/ISH negative) are excluded
      * Patients must have received prior sacituzumab govitecan and if PD-L1 ≥10% by CPS pembrolizumab with chemotherapy
   5. Classical Hodgkin Lymphoma (HL)

      * Patients must have received at least two prior systemic therapies including brentuximab vedotin (if eligible) and a prior PD-1 inhibitor
      * Patients must have experienced less than a CR (according to Lugano criteria) to anti- PD-1 treatment
   6. (Cohort 2 Dose Expansion): Non-Small Cell Lung Cancer (NSCLC)

      * Patients who have progressed after a minimum of 2 doses of a PD-1/PD-L1 treatment
      * Patients must have received prior treatment with platinum-based chemotherapy
   7. (Cohort 2 Dose Expansion) Triple Negative Breast Cancer (TNBC)

      * ER/PR and HER2 status should be defined by ASCO/CAP guidelines (JCO Allison et al 2020)
      * Patients must have received prior sacituzumab govitecan and if PD-L1 ≥10% by CPS pembrolizumab with chemotherapy
      * Patients with HER2-low tumors need to have received fam-trastuzumab deruxtecan (Enhertu)
3. Patients with NSCLC, MM, TNBC, and HNSCC must have measurable disease per RECIST 1.1. Patients with HL must have at least one measurable lesion > 1.5 cm for nodal, > 1.0 cm for extranodal FDG-avid disease by the Lugano (2014) response criteria. Tumor sites that are considered measurable must not have received prior radiation
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Adequate bone marrow function defined by absolute neutrophil (ANC) of ≥ 1.5×109/L, platelet count of ≥ 100.0×109/L, and hemoglobin of ≥ 9.0 g/dL (with or without transfusion)

   a. (Cohort 2 Dose Expansion) Adequate bone marrow function defined by absolute neutrophil (ANC) of ≥ 1.5×109/L, platelet count of ≥ 100.0×109/L, and hemoglobin of ≥ 9.0 g/dL (with or without transfusion) within 2 weeks from the first dose of CTX-8371.

   - Blood transfusion is not allowed within 2 weeks from the first dose of CTX-8371
6. Adequate hepatic function defined as serum total bilirubin ≤ 1.5 × ULN, AST/ALT ≤ 2.5 × ULN (or ≤ 5 × ULN in patients with liver metastases)
7. Adequate renal function defined as creatinine clearance ≥ 30mL/min by Cockcroft-Gault equation
8. Female patients must be surgically sterile (or have a monogamous partner who is surgically sterile) or be at least 2 years postmenopausal or commits to use 2 acceptable forms of birth control (defined as the use of an intrauterine device (IUD), a barrier method with spermicide, condoms, any form of hormonal contraceptives) or abstinence for the duration of the study and for 4 months following the last dose of study treatment. Male patients must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 4 months following the last dose of study treatment
9. Female patients who are women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening within 7 days of dosing with CTX-8371
10. Last dose of previous PD-1 or PD-L1 therapy ≥ 28 days, other anticancer therapy > 21 days (or 2 half-lives for proteins, whichever is longer), radiotherapy >21 days (concurrent localized palliative radiotherapy is allowed during CTX-8371 treatment), or surgical intervention >21 days prior to the first dose of CTX-8371
11. Resolution of all prior anti-cancer therapy toxicities ≤ Grade 2
12. Life expectancy ≥ 12 weeks
13. Capable of understanding and complying with protocol requirements
14. Signed and dated institutional review board (IRB)/independent ethics committee (IEC)-approved informed consent form (ICF) before any protocol-directed screening procedures are performed

Exclusion Criteria:

1. Developed clinically significant adverse reaction to PD-1 or PD-L1 therapy, including immune related adverse reactions, which led to discontinuation of treatment
2. Systemic therapy with immunosuppressive agents within 7 days before the start of CTX-8371 treatment. Topical, intranasal, intraocular, or inhaled corticosteroids and physiologic replacement for patients with adrenal insufficiency are allowed
3. Patient is a pregnant or lactating WOCBP
4. Prior organ transplantation
5. Patients with evidence of active hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection. Patients with positive HBsAg and/or detectable HBV DNA are eligible only if adequately controlled on antiviral therapy according to institutional standards and liver function eligibility criteria are also met. HCV patients showing sustained viral response or patients with immunity to HBV infection may enroll.
6. Active autoimmune disease or medical conditions requiring chronic steroid (i.e., > 10 mg/day prednisone or equivalent) or immunosuppressive therapy. Patients with a prior history of autoimmune disease may be eligible following discussion with the Medical Monitor
7. Other medical condition that in the opinion of the Investigator and/or Sponsor Medical Monitor may interfere with the conduct and/or interpretation of the current study, including:

   * Congestive heart failure (> New York Heart Association Class II), active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or clinically significant cardiac arrhythmias
   * QTc interval (using Fridericia correction calculation) > 480 msec
   * Known central nervous system (CNS) and brain metastasis, including asymptomatic cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Evaluate the safety and tolerability of escalating doses of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until 30 days after the last dose of CTX-8371, average of 6 months
  Number of participants with dose limiting toxicities (DLTs), treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities
Cohort 1: Determine the dose(s) of CTX-8371 to be further examined in Cohort 2 and Phase 2 studies | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks ) until 30 days after the last dose of CTX-8371 (average of 6 months )
Cohort 2: Evaluate the safety and tolerability of CTX-8371 at 3.0 mg/kg and 10.0 mg/kg | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until 30 days after the last dose of CTX-8371 (up to 2 years)
  Incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Cohort 1 and 2: Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline until confirmed disease progression (up to 2 years)
Cohort 1 and 2: Duration of Response (DOR) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (up to 2 years)
Cohort 1 and 2: Progression-Free Survival (PFS) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From first dose of CTX-8371(Cycle 1 Day 1,Cycle = 2 weeks ) until disease progression or death, whichever occur first (up to 2 years)
Cohort 1: Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as per Lugano (2014) | Baseline until confirmed disease progression (up to 2 years)
Cohort 1: Duration of Response (DOR) as per Lugano (2014) | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (up to 2 years)
Cohort 1: Progression-Free Survival (PFS) as per Lugano (2014) | From first dose of CTX-8371(Cycle 1 Day 1,Cycle = 2 weeks ) until disease progression or death, whichever occurs first
Cohort 1 and 2: Overall Survival (OS) of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1,Cycle = 2 weeks) until death (up to 2 years)
Cohort 1 and 2: Maximum serum concentration (Cmax) of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1,Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Time of maximum observed serum concentration (Tmax) of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Trough serum concentration (Ctrough) of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Area under the serum concentrations of CTX-8371 versus time curve (AUC) for CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1,Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Clearance (CL) of serum concentrations of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Volume of distribution (Vd) of serum concentrations of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Half-life (t1/2) of serum concentrations of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Dose Response for CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until treatment discontinuation
Cohort 1 and 2: Assess the immunogenicity of CTX-8371 | From first dose of CTX-8371 (Cycle 1 Day 1, Cycle = 2 weeks) until end of treatment visit
  Screen for the presence and development of antibodies against CTX-8371

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - D&H Cancer Research Center, Margate, Florida
  - Florida Cancer Specialists - Lake Nona, Orlando, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided